CLINICAL TRIAL: NCT02907827
Title: Whole-body Diffusion-weighted Magnetic Resonance Imaging and cfDNA Analysis for the Surveillance of Melanoma Patients at High Risk for Recurrence Following Surgery or Systemic Therapy
Brief Title: Whole-body DW-MRI and cfDNA Analysis for the Surveillance of Melanoma Patients at High Risk for Recurrence.
Acronym: DW-MRi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2014-BN-002
Record Dates: First submitted 2016-09-14; First posted 2016-09-20 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Melanoma
Keywords: complete remission; cfDNA; DW-MRI; surveillance
MeSH Terms: conditions — Melanoma; Pathologic Complete Response | interventions — Cell-Free Nucleic Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- stage IV melanoma CR>3years (Experimental): Stage IV: Complete remission for more than 3 years, confirmed by most recent CT or PET-CT imaging
  Interventions: Other: follow up DW MRI
- Stage III Melanoma (Experimental): AJCC Stage III: No evidence of disease on most recent CT or PET-CT imaging
  Interventions: Other: follow up DW MRI

INTERVENTIONS:
Other: follow up DW MRI — Whole-body diffusion-weighted magnetic resonance imaging and cfDNA analysis
  Other Names: cfDNA

SUMMARY:
Patients with locally advanced melanoma are at high risk for recurrence following surgical treatment. More patients with stage IV melanoma remain in complete remission following systemic therapy. No standards have been established for the surveillance of patients at high risk for recurrence. Whole-body diffusion-weighted magnetic resonance imaging and cfDNA analysis of blood are innovative imaging and laboratory investigations that may be of benefit for early detection of recurrence in this patient population.

DETAILED DESCRIPTION:
Cutaneous melanoma is the most aggressive form of skin cancer. Melanoma is the malignant cancer that originates from the melanocytes of the body (= pigmented cells of the body). Melanoma can originate from the melanocytes that are present in the skin, mucosa, or the uvea of the eye.

The incidence of melanoma is continuing to rise at a rate exceeding all other cancers. Every year approximately 132,000 and 1,000 people will be diagnosed with melanoma and 37,000 and 250 people are expected to die of the disease respectively worldwide and in Belgium. Surgical resection is curative for most cases of early identified and localized melanoma (90% long term survival for stage I disease) . Patients with stage II/III disease are at high risk of relapse after surgery, even when followed by radiotherapy and adjuvant IFN alfa-2b therapy (the risk of recurrence for these patients is 60% to 75%).

In 2010 Romano et al. published a study evaluating the time to relapse and the site of relapse in 340 patients (Figure 1: relapse free survival of all 340 patients with substages IIIA,IIIB and IIIc). Patients and/or family members discovered 62% of local and in-transit recurrences and 49% of nodal recurrences. Only 37% of patients whose first recurrence was systemic detected the recurrence themselves, either by noticing a new tumor or other symptoms that led to further evaluation. Physical examination by a physician accounted for the detection of 36% of the local and in-transit recurrences, Twenty-six percent of nodal recurrences were detected by physicians however only in 9% systemic recurrences did they discover systemic recurrence. In the remaining 63% of patients whose first detectable relapse was systemic, the relapse was asymptomatic. Radiographic tests, largely CT scans (72%), detected asymptomatic systemic relapses in 53% (n_87) of these patients. This study also demonstrated the benefit of identifying early relaps, since symptomatic relapses, as opposed to relapses discovered by physical examination or radiographic imaging, were associated with shorter survival. And confirming that a recurrence that could be completely resected was associated with longer survival (relative risk_2.31; 95% CI, 1.68 to 3.18; P_.001).

In the last several years the therapeutic landscape of melanoma has changed. The introduction of immunotherapy has increased the life expectancy for melanoma stage IV patients and even has the possibility for cure of the disease. This changes the need in screening. Since no therapeutic options were available, there was no need for a strict follow-up. The primary objective of follow-up in these patients with melanoma was to identify potentially curable locoregional recurrences and second primary cancers. Optimal follow-up strategies and intervals have not been determined, and there is no consensus. At a minimum, patients should undergo an annual routine physical examination, including a full skin assessment and palpation of the regional lymph nodes. The role of imaging in the follow-up of high risk patients is not clear. Since the introduction of newer therapies, the need for a more closer follow-up has emerged as well.

The outcome of patients with stage IV disease is grim with less than 50% of patients surviving for more than 12 months. Short-lived tumor responses are obtained in about 10-20% of patients treated with DTIC chemotherapy but no randomized trial could demonstrate a survival benefit for more complex chemotherapy regimens or so-called bio-chemotherapy regimens despite higher response rates.

In march 2011 a CTLA-4 inhibitor, Ipilimumab (Yervoy), was aproved by the FDA. It was the first treatment to prove a survival benefit in melanoma patients. An interesting aspect about the treatment with Ipilimumab is the plateau seen after 2 years.This plateau represents patient with a long term survival benefit of Ipilimumab and even the possibility of 'cure'. The patients in this population now undergo repeated imaging with PET CT and/or CT. This leads to a high radiation burden for this patients. The DW-MRI could in this population have a benefit.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignant melanoma;
* AJCC Stage III: No evidence of disease on most recent CT or PET-CT imaging
* Stage IV: Complete remission for more than 3 years, confirmed by most recent CT or PET-CT imaging

Exclusion Criteria:

* Contra-indication for MRI: pacemaker, metallic foreign body in eye, recent operation with prosthetic material (< 6weken)
* Claustrophobia
* Metallic devices implanted such as hip prostheses, since this can alter the imaging quality

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-11; Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
explorative evaluation of the use of DWMRI in the follow-up of high risk melanoma patients | 5years

SECONDARY OUTCOMES:
• Distant metastasis-free survival (for stage III patients only), overall survival | 5years
• Registration of the nature and result of salvage therapies offered at the time of detection of recurrence/progression | 5 years
• Explore the correlation of cfDNA measurements and the clinical or MRI based diagnosis of recurrence/progression | 5years

CONTACTS AND LOCATIONS:
Overall Officials: Bart Neyns, Md Phd, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (2):
- Belgium (2):
  - UZ Brussel, Jette, Brabant
  - UZ Brussel, Brussels

IPD SHARING:
Plan to Share IPD: Yes
anonymous